CLINICAL TRIAL: NCT00109538
Title: A Pivotal Randomized Study of Lonafarnib Versus Placebo in the Treatment of Subjects With Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) Who Are Platelet Transfusion Dependent With or Without Anemia
Brief Title: Study of Lonafarnib Versus Placebo in Subjects With Either Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) (Study P02978AM3)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P02978
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Myelodysplasia; Myelomonocytic
Keywords: Lonafarnib
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts | interventions — lonafarnib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lonafarnib (Experimental): Lonafarnib 200 mg twice daily, oral, continuously
  Interventions: Drug: Lonafarnib
- Placebo (Placebo Comparator): Placebo, BID, oral
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lonafarnib — 200 mg twice daily (BID, ie, approximately 12 hours apart with food), oral, continuously, or until unacceptable toxicity or transformation to AML, or disease progression, or other discontinuation criteria
  Other Names: SCH 66336
  Arms: Lonafarnib
Other: Placebo — BID, oral, continuously, or until unacceptable toxicity or transformation to AML, or disease progression, or other discontinuation criteria
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the benefit of lonafarnib (versus placebo) in patients with myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML). Benefit will be measured by achievement of platelet transfusion independence for at least 8-consecutive weeks, and without simultaneous worsening of hemoglobin and/or need for red blood cell (RBC) transfusion. Additional endpoints will be hematologic response (which includes complete remission, partial remission, hematologic improvement), number of RBC transfusions, bleeding events, infections and safety.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MDS (RA, RARS, RAEB, RAEB-T) or CMML according to FAB classification.
* Platelet transfusion dependence (requiring 1 to 8 platelet transfusion events every 4 week period (Day 84 to Day 57, Day 56 to Day 29, and Day 28 to Day 1) over an 8-week retrospective and 4-week prospective screening period).
* The individual number of platelet transfusion events during the three 4-weekly periods (Day 84 to Day -57; Day -56 to Day 29; Day -28 to Day -1) must not differ by greater more than 2 from the average number of platelet transfusion events during the 12 week screening period.
* If the subject is RBC transfusion dependent, the number of RBC transfusion events during the three 4-weekly periods (Days -84 to -57; Day -56 to Day 29 and Day -28 to Day -1) must not differ by more than 2 from the average number of RBC transfusion events during this 12 week screening period.

ECOG PS 0-2.

Exclusion Criteria:

* Subjects with chemotherapy/radiotherapy-associated secondary MDS.
* <12 Weeks (prior to Day-1 Randomization) from any investigational drug use, any chemotherapy, radiotherapy, immunotherapy and any other treatment or MDS/CMML other than best supportive care.
* Hx of bone-marrow or peripheral stem-cell transplantation or treatment with donor lymphocyte infusion.
* Hx of AML.
* Known hx of immune thrombocytopenic purpura.
* Marked baseline prolongation of QTc interval, CTCAE Grade >=1.
* Use of ketokonazole within 72 hours prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieved platelet transfusion independence for any 8-consecutive week period after randomization without worsening of RBC transfusion requirements or hemoglobin (untransfused) during the same 8-consecutive-week period. | Any 8-consecutive week period after randomization

SECONDARY OUTCOMES:
Hematologic response rate (CR, PR, HI), number of RBC transfusion events during a 4-week period, active bleeding events (number and severity), number of CTCAE Grade 3 and 4 infections and days of acute intervention, and safety. | Any 8-consecutive week period after randomization